CLINICAL TRIAL: NCT06343025
Title: The Effect of Different Exercise Programs on Glycemic Control, Body Composition, Balance and Physical Activity Level in Individuals With Prediabetes
Brief Title: The Effects of Tai Chi and Pilates for Individuals With Prediabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: Hasan Kalyoncu University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hasan Kalyoncu University
Record Dates: First submitted 2024-03-27; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: PreDiabetes
Keywords: prediabetes; Tai Chi; Pilates; Exercise
MeSH Terms: conditions — Prediabetic State; Motor Activity

STUDY DESIGN:
Intervention Model Description: Individuals will be divided into 3 groups: Clinical Pilates group, Tai Chi group and Control group. 3 groups. 3 groups will be measured at the same time and then the exercise part will begin.
Who Masked: Outcomes Assessor
Masking Description: Outcomes ,Assesor, who will make the evaluations in the first week and after 12 weeks, will not know which group the people are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pilates Group (Experimental): Individuals will perform clinical pilates exercises for 60 minutes, 3 days a week for 12 weeks. It includes 45 minutes of basic pilates exercises, 10 minutes of warm-up and 5 minutes of cool-down exercises. In addition, Diet will be recommended by the doctor as routine treatment.
  Interventions: Other: Pilates Exercises Group
- Tai Chi Group (Experimental): Individuals will perform Tai Chi exercises for 60 minutes, 3 days a week for 12 weeks. It includes 45 minutes of Tai Chi movements, 10 minutes of warm-up and 5 minutes of cool-down exercises. In addition, Diet will be recommended by the doctor as routine treatment.
  Interventions: Other: Tai Chi Exercises Group
- Control Group (No Intervention): The control group will not be given any training. Diet and brisk walking 3 days a week will be recommended by the doctor as routine treatment for the control group.

INTERVENTIONS:
Other: Pilates Exercises Group — Individuals will perform clinical pilates exercises for 60 minutes, 3 days a week for 12 weeks. It includes 45 minutes of basic pilates exercises, 10 minutes of warm-up and 5 minutes of cool-down exercises.
  Arms: Pilates Group
Other: Tai Chi Exercises Group — Individuals will perform Tai Chi exercises for 60 minutes, 3 days a week for 12 weeks. It includes 45 minutes of Tai Chi movements, 10 minutes of warm-up and 5 minutes of cool-down exercises.
  Arms: Tai Chi Group

SUMMARY:
The purpose of this study; To investigate the effects of Clinical Pilates and Tai Chi exercises on glycemic control, body composition, balance function and physical activity level in individuals with prediabetes.

DETAILED DESCRIPTION:
The purpose of this study; To investigate the effects of Clinical Pilates and Tai Chi exercises on glycemic control, body composition, balance function and physical activity level in individuals with prediabetes. Method: 54 individuals diagnosed with Prediabetes in the Endocrinology and Metabolic Diseases Polyclinic at Niğde Ömer Halisdemir Training and Research Hospital will participate in our study. Individuals will be divided into 3 groups: Clinical Pilates group, Tai Chi group and control group. Before exercise, routine blood tests of individuals will be performed and their fasting and postprandial blood glucose and HbA1C (Glycosized Hemoglobin) levels will be checked. Bioelectrical Impedance Device will be used to evaluate body composition. Timed Up and Go Test and Berg Balance Scale will be used to evaluate individuals' balance functions. Physical Activity level of individuals will be measured using the International Physical Activity Level Scale (IPAQ) and the Accelerometer device. Evaluations will be repeated in all groups at the end of the 12-week exercise application. SPSS (Statistical Package Program for Social Science) software will be used to analyze the data. Statistical analysis of the study will be done with Wilcoxon related two-sample test for intra-group measurements, and Man Whitney U test for inter-group evaluations. For the significance level, p value will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent biochemistry analysis for their glycemic control as part of routine checks at the Endocrinology and Metabolic Diseases Polyclinic.
* Patients who do not use any medication related to prediabetes
* Being able to walk independently
* Volunteering to exercise at least 3 days a week within the scope of the research

Exclusion Criteria:

* Those diagnosed with type 1 diabetes, Latent Autoimmune Diabetes in Adults (LADA)
* Going into a diabetic ketoacidosis coma,
* Having an orthopedic problem that prevents walking and exercising
* Having an orthopedic or vascular problem with the foot
* Having any neurological disease
* Cardiac, pulmonary or systemic disease that would prevent exercise have
* Losing more than 4 kg of weight per month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Glisemic Control | 2024- 2025
  In our study, Hemoglobin A1C (HbA1C), fasting blood glucose and postprandial blood glucose values will be examined from routine biochemistry analyses.
Body Composition | 2024-2025
  In our study, the body composition of the participants will be evaluated using the Bioelectrical Impedance Device.
Balance | 2024-2025
  In our study, it was decided to use Berg Balance Scale and Timed Up and Go Test to measure balance.
Physical Activity Level | 2024-2025
  In our study, the International Physical Activity Scale (IPAQ) and Accelerometer will be used to determine the physical activity level.